CLINICAL TRIAL: NCT04753463
Title: Assessment of the Impact of COVID-19 Pandemic on Residents Training and Mental Health in Poland
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: 1775
Record Dates: First submitted 2021-02-04; First posted 2021-02-15 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2
Keywords: Residents training
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residents of Ophthalmology working on COVID-19 departments: Residents of ophthalmology working on COVID-19 departments and dealing with SARS-CoV-2 positive patients
  Interventions: Other: Survey
- Residents of Ophthalmology working on general ophthalmic departments: Residents of Ophthalmology working on general ophthalmic departments and not dealing with SARS-CoV-2 positive patients
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The on-line questionnaire which assess the subjective feelings of residents of pandemic impact on ophthalmology training programs

SUMMARY:
The aim of study is to investigate the impact of SARS-CoV-2 on ophthalmology training programs among residents. To the best of our knowledge this study is the first of its kind in Poland. The impact of COVID-19 on ophthalmology training programs is largely unknown as there are only few studies assessing the above issue from the resident's point of view.

DETAILED DESCRIPTION:
The novel coronavirus SARS-CoV-2, responsible for Coronavirus Disease 2019 (COVID-19), was first identified at the end of the year 2019 in Wuhan (China). A rapid spread of the disease resulted in global threat to public health. On 11 March 2020 the World Health Organization (WHO) announced the state of pandemic. In Poland, the first confirmed case of COVID-19 was reported on 4 March 2020 and subsequent growing number of patients has placed tremendous strain on healthcare system. The crisis situation prompted immediate action to divert healthcare resources for the treatment of patients with COVID-19 and to limit the spread of the infection. In accordance with the decision of the Minister of Health of March 13th, 2020, more than twenty hospitals were established to admit only the SARS-CoV-2 affected patients. Moreover, all hospitals were recommended to limit their planned activity and to perform only urgent and emergency services.

The investigators hypothesize that those changes in healthcare system and restrictions established in public area during pandemic caused significant difficulties in residency training considering clinical and surgical practice as well as didactic activities. In spite of gradual reopening the routine services over the last few months, social distancing rules are still in force. Accordingly, different methods of virtual teaching were introduced including, inter alia, organisation of courses, lectures and conferences in form of on-line meetings.

The aim of current study is to investigate the impact of SARS-CoV-2 on ophthalmology training programs among residents. To the best of our knowledge this study is the first of its kind in Poland. The impact of COVID-19 on ophthalmology training programs is largely unknown as there are only few studies assessing the above issue from the resident's point of view.

The investigators believe that this investigations will address this gap in the literature and could be used to initiate the new solutions in order to maintain successful residency training during pandemic. Opinions regarding the efficiency of e-learning methods and on-line meetings may be crucial to innovate the conventional teaching way permanently in the future.

ELIGIBILITY:
Inclusion Criteria:

* male and female in the age of 25-35 during residence training

Exclusion Criteria:

* lack of consent for participating in survey

Ages: 25 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Residents of ophthalmology (male and female), in the age of 25-35 working on ophthalmology departments
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
questionnaire assessing the incidence of disturbance of COVID-19 pandemic on ophthalmology training programs among residents | 1 month
  the opinion of ophthalmology training programs among residents assessed with the questionnaire collecting demographics (age, gender), domicile (state, union territory), current professional status (in training or practising), type of practice (solo, group, institutional, governmental, non-governmental), marital status (married, single), impact of COVID-19 on their training or ophthalmology practice, and impact on income and ability to meet living expense

SECONDARY OUTCOMES:
questionnaire assessing the negative impact of COVID-19 pandemic on mental health among ophthalmology residents | 1 month
  the opinion on impact for mental health among residents assessed with the Patient Health Questionnaire-9 (PHQ-9). PHQ-9 is a selfreport measure that is used to assess the severity of depression over the prior 2 weeks. Response to the nine questions are graded as 0 (not at all), 1 (several days), 2 (more than half the days), and 3 (nearly every day). The total score of PHQ-9 that categorizes depression is as follows: minimal/no depression (0-4), mild depression (5-9), moderate depression (10-14), or severe depression (15-21).
questionnaire assessing the attitude on COVID-19 vaccination of ophthalmology residents | 1 month
  the attitude towards the vaccination against the SARS-CoV-2 among residents assessed with the questionnaire with open questions about the willingness of taking the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Marek MD Rękas, Prof, Study Chair — Wojskowy Instytut Medyczny
Locations (2):
- Poland (2):
  - Medical University, Bialystok
  - Ophthalmology Clinic Medical University of Bialystok, Bialystok

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that underlie the results reported in this article are available upon reasonable request for academic and non-commercial purposes beginning with article publication and ending 5 years thereafter. Proposals should be submitted to joannakonopinska@o2.pl for review and approval by an internal steering committee. Qualified researchers with reasonable proposals will be provided access to the data along with the redacted study protocol and statistical analysis plan to achieve the specified aims in their approved proposal after signing a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Since the time of publication up to 5 years
Access Criteria: As above

REFERENCES:
- [Result] Silva N, Laiginhas R, Meireles A, Barbosa Breda J. Impact of the COVID-19 Pandemic on Ophthalmology Residency Training in Portugal. Acta Med Port. 2020 Oct 1;33(10):640-648. doi: 10.20344/amp.14341. Epub 2020 Sep 10. PMID 32914750
- [Result] Mishra D, Nair AG, Gandhi RA, Gogate PJ, Mathur S, Bhushan P, Srivastav T, Singh H, Sinha BP, Singh MK. The impact of COVID-19 related lockdown on ophthalmology training programs in India - Outcomes of a survey. Indian J Ophthalmol. 2020 Jun;68(6):999-1004. doi: 10.4103/ijo.IJO_1067_20. PMID 32461413
- [Result] El-Saied HMA, Salah Eddin Abdelhakim MA. Impact of COVID-19 Pandemic on Young Ophthalmologists in Cairo University Hospitals. Semin Ophthalmol. 2020 Aug 17;35(5-6):296-306. doi: 10.1080/08820538.2020.1826046. Epub 2020 Oct 5. PMID 33017198